CLINICAL TRIAL: NCT02591654
Title: A Feasibility Study of MRI and PET Imaging to Assess Response to MK-3475 (Pembrolizumab) in Patients With Metastatic Melanoma
Brief Title: MRI and PET to Assess Pembrolizumab Response
Acronym: MPAK
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Columbia University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAO2558
Record Dates: First submitted 2015-10-21; First posted 2015-10-29 (Estimated); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Malignant Melanoma, Metastatic
Keywords: FLT; Pembrolizumab; Metastatic Melanoma; MK-3475
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — pembrolizumab; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab and FLT (Experimental): Subjects will receive WB-DW MRI and FLT PET to assess disease burden after receiving pembrolizumab.
  Interventions: Drug: Pembrolizumab; Drug: FLT PET

INTERVENTIONS:
Drug: Pembrolizumab — Each patient will receive pembrolizumab 200mg administered as a 30 minute intravenous (IV) infusion every 3 weeks for an indefinite period.
  Other Names: MK-3475
Drug: FLT PET — FLT PET/CT is increasingly being utilized as an early PD biomarker in cancer given the close association between FLT uptake and proliferative index.
  Other Names: [18F]-fluorothymidine (FLT) PET

SUMMARY:
The purpose of this study is to test two imaging techniques, one called whole body (WB) diffusion weighted (DWI) magnetic resonance imaging (MRI) (WB-DWI MRI), and another called Fluorine-18 3'-deoxy-3'-fluorothymidine positron emission tomography (PET) (F-18-FLT PET). The goal is to see whether these imaging techniques would allow the study doctors to see changes in the size of a tumor earlier for patients with metastatic melanoma receiving Pembrolizumab (MK-3475).

DETAILED DESCRIPTION:
There is a growing body of evidence that demonstrates that tumor proliferation, measured classically by immunohistochemical evidence of increased Ki-67 expression, can be reliably determined in vivo using radiolabeled thymidine. The development of [18F]-fluorothymidine (FLT) PET has been reliably identified as a marker of cellular proliferation, and has been shown to identify changes in proliferation in successfully treated patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of melanoma
* Stage III or stage IV metastatic melanoma
* Disease that is measurable. This is defined as lesions measuring at least 10mm on radiologic imaging. For lymph node disease, the lesion must measure at least 15 mm or have been biopsied and shown to contain melanoma. Skin or mucosal lesions that are not measurable on radiologic imaging but measure at least 10mm on clinical exam are also acceptable. (See Section 13.2 for detailed definition of measurable disease)
* Disease is termed unresectable or the patient refuses resection
* The Eastern Cooperative Oncology Group (ECOG) performance status of 1 or better
* Age ≥18 years. This is due to the limited data with pembrolizumab in children younger than 18 years of age.
* Normal organ and marrow function as defined below

  * Aspartate aminotransferase (AST) (SGOT) or alanine aminotransferase (ALT) (SGPT) ≤2.5 × institutional upper limit of normal (≤5 x upper limit of normal for patient with liver metastasis)
  * Total bilirubin within 1.5 x institutional level of normal or direct bilirubin ≤ upper limit of normal (ULN) for patient with total bilirubin levels > 1.5 ULN)
  * Hemoglobin ≥ 9.0g/dL or ≥5.6mmol/L
  * Absolute neutrophil count ≥1,000/microliters (mcL)
  * Platelets ≥ 75,000/mcL
* The effects of pembrolizumab on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of pembrolizumab administration.
* Women of child-bearing potential must have a negative urinary or serum pregnancy test.

Exclusion Criteria:

* Prior therapy with anti-PD-1 antibody
* The patient has symptomatic brain metastases. Asymptomatic brain metastases are permitted provided that there is no steroid requirement, no more than 4 metastases detected on standard MRI imaging, no metastatic brain lesion that is > 3 cm in size, and no lepto-meningeal disease.
* Patient has not recovered to Grade 0-1 from adverse events due to prior chemotherapy, radiation, or biological cancer therapy (including monoclonal antibody (mAb)).
* The patient is not recovered from minor or major surgery and is less than 4 weeks from major surgery prior to starting treatment with pembrolizumab
* Significant auto-immune disease requiring hospitalization within the past two years or any history of life-threatening auto-immune disease
* Immunosuppressive therapy including systemic corticosteroids except for maintenance dosing for adrenal insufficiency
* Concurrent use of any other investigational agents
* Active central nervous system metastasis and/or carcinomatous meningitis causing symptoms.
* Known additional malignancy that is progressing or requires active treatment with the exceptions of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Active autoimmune disease or a syndrome that requires systemic steroids or immunosuppressive agents with the exceptions of replacement dose steroids for adrenal insufficiency, vitiligo, resolved childhood asthma/atopy, intermittent use of inhaled steroids, local steroid injections, hypothyroidism stable on hormone replacement, and Sjogren's syndrome
* Active tuberculosis
* Hypersensitivity to pembrolizumab or any of its excipients.
* Expected to require any other form of systemic antineoplastic therapy while receiving pembrolizumab
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, autoimmune diseases, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with a pacemaker, stainless steel aneurysm clip or any other magnetic resonance (MR) contraindicated implant or foreign body would warrant exclusion from this study. Pacemakers may be reprogrammed or turned off by the strong MRI magnetic field. Radio-frequency (RF) fields in MR can also cause severe heating of pacemaker lead tips. Steel aneurysm clips are prone to torque in the strong MR field which can displace the clips and may damage the vessel, resulting in hemorrhage, and/or death.
* All patients and volunteers are screened before MR examination using a MRI safety screening Questionnaire as part of the New York Presbyterian/Columbia University Medical Center (NYP/CUMC) MRI safety policy. Any patient who would normally be excluded by this screening process would also be excluded from this study.
* Pregnant or breastfeeding women are excluded from this study because of the unknown effects of the study agent on the unborn child and the possible adverse impact of immune activation on pregnancy. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pembrolizumab breastfeeding should be discontinued if the mother is treated with pembrolizumab.
* Male who is expecting to father a child during the treatment period.
* History of pneumonitis requiring hospitalization or systemic immune suppressive therapy.
* Significant immunodeficiency making the patient unlikely to benefit from pembrolizumab therapy including a diagnosis of acquired immune deficiency syndrome (AIDS), active hepatitis B or hepatitis C, or organ transplant requiring immunosuppressive therapy.
* Received a live virus vaccine within 30 days of planned start of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2022-10 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of lesion detection (sensitivity) | Baseline
  Sensitivity of WB-DW MRI and FLT-PET imaging in lesion detection and evaluation for metastatic melanoma.

SECONDARY OUTCOMES:
Difference in lesion metrics | Baseline, 2 years
  Lesion metrics including diameter and intensity as measured by FLT-PET and WB-DWI MRI will be compared with standard RECIST and volumetric criteria as well as Immune Response Criteria (IRC).
Change in patient response (immunoscore) | Baseline, 2 years
  Assessed by programmed cell death protein 1 (PD-1), programmed death-ligand 1 (PD-L1), and programmed death-ligand 2 (PD-L2) expression, quantification of infiltrating cluster of differentiation 8 (CD8+) T cells at the invasive margin and within the center of the tumor, and assessment of cluster of differentiation 2 (CD2) expression. Formalin fixed paraffin embedded sections will be used. Cluster of differentiation 3 (CD3) and CD8 will be stained for and the immunoscore will be calculated using standard methods.
Change in patient response (expression levels) | Baseline, 2 years
  Assessed by NanoString with measurement of immune related genes. Expression levels will be compared pre-treatment and post-treatment.
Change in RECIST Index | Baseline, 6 weeks
  Index lesions identified on the baseline standard Response Evaluation Criteria In Solid Tumors (RECIST) image set will be evaluated for changes in FLT maximum standardized uptake value (SUVmax) and standardized uptake volume (SUVvol), and changes in antibody-drug conjugate (ADC) on DWI MRI at 6 weeks compared with baseline. These early response measures will then be compared with RECIST response measurements on conventional imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Saenger, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center / NewYork-Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Herbert Irving Comprehensive Cancer Center — http://www.hiccc.columbia.edu